CLINICAL TRIAL: NCT05831358
Title: Early Detection of Multiple Myeloma to Fight Cancer Disparities: A Screening and Patient Navigation Program
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CASE1A23
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma; Monoclonal Gammopathy of Undetermined Significance; Smoldering Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma; Monoclonal Gammopathy of Undetermined Significance; Smoldering Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Not a randomized trial; use of convenience sampling.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multiple Myeloma Screening Experience (Experimental): Participants will partake in a multiple myeloma screening program. The screening involves a blood sample and the completion of a questionnaire to gauge participants' multiple myeloma knowledge.
  Interventions: Other: Multiple Myeloma M-Protein Analysis; Other: Multiple Myeloma Knowledge Questionnaires

INTERVENTIONS:
Other: Multiple Myeloma M-Protein Analysis — Participants will be screened with a blood test for monoclonal protein analysis
Other: Multiple Myeloma Knowledge Questionnaires — Participants will complete two questionnaires to share their attitudes toward their screening experience and completion of knowledge questions to gauge community reception and participant multiple myeloma knowledge.

SUMMARY:
This project will pilot the expansion of the existing Taussig Outreach Program's community outreach and patient navigation model to study the multiple myeloma (MM) screening program. This involves analyzing community reception, screening program methods, reasons patients decided to participate, reasons patients declined participation, and participant views and attitudes. This study also aims to gauge the current and general understanding of MM. This study seeks to recruit participants in the pilot screening program to promote early detection. Participants who have abnormal results will receive patient navigation for further diagnostics and testing.

DETAILED DESCRIPTION:
Multiple Myeloma (MM) is a hematologic cancer of antibody-producing plasma cells. Multiple Myeloma is always preceded by a pre-malignant condition called monoclonal gammopathy of undetermined significance (MGUS) or smoldering multiple myeloma. Despite multiple therapeutic advances, there remains no cure for multiple myeloma. The disease is treated and monitored throughout a person's lifetime. This is why screening for early detection of this disease is important; however, MGUS and smoldering multiple myeloma are only diagnosed when they are found incidentally on labs during tests for unrelated symptoms. There are no current universal screening guidelines for MM. Among those who may benefit from MM screenings include African American/Black individuals, as it is twice as common in this population compared to Caucasian/White individuals. This study aims to develop a screening program specifically targeting underserved African American/Black individuals. This project will expand the existing Taussig Community Outreach screening program to include screening for multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Participant self-identifying as, or perceived as, Black and/or African-American
* 50 years of age or older

Exclusion Criteria:

* Participants who do not self-identify as Black and/or African American
* Under the age of 50 years

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2023-06-16 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
To conduct and evaluate a study that incorporates patient navigation programs to recruit and screen participants for Multiple Myeloma and its disease precursors, MGUS or smoldering MM | 12 months
  The goal is to leverage the existing model of community outreach and patient navigation to study the MM screening program, including community reception, screening program methods, reasons patients decided to participate, reasons patients declined participation, and participant views and attitudes. This will be measured by the overall community reception of this screening being offered.
To conduct and evaluate a study that incorporates patient navigation programs to recruit and screen participants for Multiple Myeloma and its disease precursors, MGUS or smoldering MM | 12 months
  The goal is to leverage the existing model of community outreach and patient navigation to study the MM screening program, including community reception, screening program methods, reasons patients decided to participate, reasons patients declined participation, and participant views and attitudes. This will be measured by participant questionnaires detailing their attitudes toward, and experience, of the screening.
To study participant knowledge of Multiple Myeloma | 12 months
  Participants will gain knowledge about Multiple Myeloma from the time of the screening to the time of follow-up one week or more after the screening. This will be measured by examining the difference in participant post-screening questionnaire results.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Valent, MD, Principal Investigator — Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No